CLINICAL TRIAL: NCT01670838
Title: Cardiopulmonary Complication in Aneurysmal Subarachnoid Haemorrhage Patients
Acronym: SAHHEART
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Maarit Lang, MD, Kuopio University Hospital
Other Study IDs: Kuopio UH
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Aneurysmal Subarachnoid Heamorrhage; Nontraumatic Subarachnoid Haemorrhage
Keywords: subarachnoid haemorrhage; cardiopulmonary complications
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MICRORNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subarachnoid haemorrhage: nontraumatic subarachnoid haemorrhage

SUMMARY:
This is a prospective cohort study investigating cardiac function and cardiac biomarkers in patients with acute Aneurysmal Subarachnoid Haemorrhage (aSAH). The aims of the study are to document the incidence of myocardial dysfunction,to find the predictive factors of myocardial dysfunction, describe heart rate variability and to assess the impact of all cardiac problems on morbidity and mortality.

DETAILED DESCRIPTION:
Laboratory markers daily: Routine laboratory test (blood gases, haemoglobin, thrombocytes, leukocytes, INR, bilirubin, creatinine, c-reactive protein, CK, CK-MB, Tnt, BNP, sodium, potassium, magnesium) are taken at 8 a.m. Study laboratory tests (sensitive ischemia markers, remodelling marker MMP-9 and CgA as surrogate marker for increased sympathetic activity) are taken four times during study period at the same time as cardiac ECHOes and Holtering. Gene sample is taken once on day one.

Primary outcome measurement is to document the incidence of myocardial dysfunction and the predictive factors during the hospital stay and at three months.

Secondary outcome is to assess the impact of cardiac problems on morbidity and mortality during first three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nontraumatic subarachnoid haemorrhage
* Age > 18 years
* Aneurysmal bleeding

Exclusion Criteria:

* No consent
* Age < 18 years
* Anticipated brain death < 24 hours
* Otherwise moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study material consists of 200 consecutive aSAH-patients treated in Kuopio University Hospital and Turku University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac failure and the impact of cardiac problems on morbidity | 6 months
  The aims of the study are:
  1. to document the incidence of myocardial dysfunction
  2. to find the predictive factors of myocardial dysfunction as determined by the severity aneurysmal bleeding (Hunt and Hess-grading, Glasgow coma score, Fisher scale) and demographic factors
  3. to find predictive factors for myocardial dysfunction as determined by laboratory findings, electrocardiography, and echocardiography
  4. to describe heart rate variability
  5. to assess the impact of all cardiac problems on morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Stepani Bendel, PhD, MD, Study Director — Senior consultant, intensivist; Maarit Lång, MD, Principal Investigator — Senior consultant, intensivist
Locations (3):
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No